CLINICAL TRIAL: NCT06015737
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled, Phase III Study to Evaluate the Efficacy and Safety of Anifrolumab in Adults With Chronic and/or Subacute Cutaneous Lupus Erythematosus Who Are Refractory and/or Intolerant to Antimalarial Therapy.
Brief Title: A Phase III Study to Investigate the Efficacy and Safety of Anifrolumab in Adults With Chronic and/or Subacute Cutaneous Lupus Erythematosus
Acronym: LAVENDER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D346BC00001; 2021-003698-70 (EudraCT Number)
Record Dates: First submitted 2023-08-01; First posted 2023-08-29 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Cutaneous Lupus Erythematosus
Keywords: Lupus erythematosus; Cutaneous lupus erythematosus; Anifrolumab; Cutaneous Lupus Erythematosus Disease Area Severity Index; Subacute lupus; Discoid lupus
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Discoid | interventions — anifrolumab

STUDY DESIGN:
Intervention Model Description: This is a parallel group treatment study with two arms.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anifrolumab (Experimental): Participants will receive anifrolumab as a SC injection from Week 0/Day 1 up to Week 51.
  Interventions: Combination Product: Anifrolumab
- Placebo (Placebo Comparator): Participants will receive placebo as a SC injection from Week 0/Day 1 up to Week 23. From Week 24 the participants will receive anifrolumab up to and including Week 51.
  Interventions: Other: Placebo

INTERVENTIONS:
Combination Product: Anifrolumab — Anifrolumab will be provided as a solution for injection in accessorized pre-filled syringe (aPFS).
  Arms: Anifrolumab
Other: Placebo — Matching placebo solution for injection in aPFS.
  Arms: Placebo

SUMMARY:
This study aims to evaluate the efficacy and safety of subcutaneous (SC) anifrolumab versus placebo in adult participants with chronic and/or subacute cutaneous lupus erythematosus (CLE).

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, Phase III study to evaluate the efficacy and safety of anifrolumab in adults with chronic and/or subacute CLE who are refractory and/or intolerant to antimalarial therapy. The study has a randomized, 24-week double-blind, placebo-controlled study period (Week 0 to Week 23), to evaluate the efficacy and safety of anifrolumab. The double-blind study period will be followed by an open-label, uncontrolled treatment period in which all participants will receive treatment with anifrolumab from Week 24 to Week 51. After the open-label treatment period, participants will enter a 12-week Safety Follow-up Period.

ELIGIBILITY:
Key inclusion criteria:

* Participants must have a confirmed diagnosis of CLE. Diagnosis must be clinically and histologically confirmed with the following:

  * CLASI-A total score ≥ 10 points at Screening and confirmed at randomization.
  * Inadequate response or intolerant to antimalarial therapy.
* Participants should have no medical history or signs or symptoms of active or prior tuberculosis infection (TB) and the same should reflect in chest radiograph or a chest CT scan result.
* Contraceptive use by males and females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Key exclusion criteria:

* History or evidence of suicidal ideation.
* Severe or life-threatening Systemic lupus erythematosus (SLE).
* Active SLE or Sjögren's Syndrome.
* Any active skin conditions other than CLE that may interfere with the study.
* History of, or current diagnosis of, catastrophic antiphospholipid syndrome (APS).
* History of recurrent infection requiring hospitalization and IV antibiotics.
* COVID-19 infection.
* Any history of an anaphylactic reaction to human proteins, or monoclonal antibodies.
* At screening, if participants do not meet the eligibility criteria assessed based on laboratory test results e.g tests for total bilirubin, serum creatinine etc.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2024-06-29 (Actual); Primary Completion 2026-11-13 (Estimated); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a 70% reduction relative to baseline in the Cutaneous Lupus Erythematosus Disease Area and Severity Index-Activity (CLASI-A) score | At Week 24
  The CLASI is a validated index used for assessing the cutaneous lesions of SLE. It consists of 2 separate scores: i) activity of the disease, and ii) measure of damage. The CLASI instrument will be used at each study visit to capture individual skin manifestation scores. CLASI-70 responder (Yes/No) is defined as a participant who achieves a 70% reduction relative to baseline in CLASI-A score. Otherwise, the participant is considered a non-responder.

SECONDARY OUTCOMES:
Change from baseline in total CLASI-A score | At Week 24
  The CLASI-A is a validated index used for assessing the cutaneous lesions of SLE.
Number of participants with CLASI-70 response | At Week 12
  The CLASI is a validated index used for assessing the cutaneous lesions of SLE. CLASI-70 responder is defined as a participant who achieves a 70% reduction relative to baseline in CLASI-A score. Otherwise, the participant is considered a non-responder.
Number of participants with ≥ 7-point reduction from baseline in CLASI-A total score | At Week 12
  The CLASI is a validated index used for assessing the cutaneous lesions of SLE. A 7-point reduction CLASI-A is established as clinically meaningful improvement in disease for CLE and as being impactful for patients.
Number of participants with CLASI-50 response | At Week 12 and Week 24
  The CLASI is a validated index used for assessing the cutaneous lesions of SLE. CLASI-50 responder is defined as a responder (yes/no) is defined as a participant who achieves at least a 50% reduction relative to baseline in CLASI-A score. Otherwise, the participant is a non-responder.
Number of participants who are sustained CLASI-70 responders | Up to Week 52
  The CLASI is a validated index used for assessing the cutaneous lesions of SLE. CLASI-70 responder is defined as a participant who achieves a 70% reduction relative to baseline in CLASI-A score. Otherwise, the participant is considered a non-responder. Amongst participants randomized to anifrolumab, the number of participants who maintained a CLASI-70 response from Week 24 up to Week 52 will be evaluated.
Serum trough (pre-dose) concentrations of anifrolumab | Double-blind: Pre-dose on Day 1 (Week 0), Weeks 1, 4, 12, 24; Open-label: Weeks 40, and 52 or early discontinuation visit [EDV] and follow-up visit (13 Weeks after last dose)
  The Ctrough of subcutaneously administered anifrolumab in participants with chronic and/or subacute CLE will be evaluated.
Number of participants with positive antidrug antibody | Double-blind: Pre-dose on Day 1 (Week 0), Weeks 4, 12, and 24; Open-label: Pre-dose on Weeks 40, and 52 or EDV and follow-up visit (13 weeks after last dose)
  The immunogenicity of subcutaneously administered anifrolumab in participants with chronic and/or subacute CLE will be evaluated.
Percent change from baseline in suppression of the Interferon 21-gene | Double-blind: Day 1 (Week 0), Week 1, 4, 12, and 24; Open-label; Week 40 and 52 or EDV and follow-up visit (13 weeks after last dose)
  The pharmacodynamics of subcutaneously administered anifrolumab in participants with chronic and/or subacute CLE will be evaluated.
Change from baseline in Skindex-29+3 Symptom domain scores | At Week 24
  The Skindex-29+3 is based on a previous instrument, the Skindex-29 and has been modified to include items related to CLE. The instrument consists of 33 items, which are used to calculate 4 domains: Symptoms (7 items), Emotions (10 items), Functioning (12 items), and Lupus-specific (3 items). The remaining item asks the participants to rate how often they worry about side effects from treatment; however, this item is not used to calculate the domain scores. The response options are on a 5-point verbal rating scale, ranging from 1 (Never) to 5 (All the time). The instrument has a recall period of the previous 4 weeks. Each domain score ranges from 0 to 100 points, with higher scores indicating worse health-related quality of life.
Change from baseline in Skindex-29+3 Emotion domain scores | At Week 24
  The Skindex-29+3 is based on a previous instrument, the Skindex-29 and has been modified to include items related to CLE.
Change from baseline in Skindex-29+3 Function domain scores | At Week 24
  The Skindex-29+3 is based on a previous instrument, the Skindex-29 and has been modified to include items related to CLE.
Change from baseline in Skindex-29+3 Lupus-Specific domain scores | At Week 24
  The Skindex-29+3 is based on a previous instrument, the Skindex-29 and has been modified to include items related to CLE.
Change from baseline in Skindex-29+3 Total score | At Week 24
  The Skindex-29+3 is based on a previous instrument, the Skindex-29 and has been modified to include items related to CLE.
Time from IP start date to CLASI-70 response. | From Week 0/Day 1 up to Week 24
  To assess the efficacy of anifrolumab compared with placebo on the onset of reduction in skin manifestations in participants with chronic and/or subacute CLE.
Time from IP start date to CLASI-50 response. | From Week 0/Day 1 up to Week 24
  To assess the efficacy of anifrolumab compared with placebo on the onset of reduction in skin manifestations in participants with chronic and/or subacute CLE.

OTHER OUTCOMES:
Number of participants with adverse events | Screening (up to and including 42 days before Day 1) until Safety Follow-up Period (12 weeks from Week 52/EDV)
  To evaluate the safety and tolerability of anifrolumab compared with placebo in participants with CLE.

CONTACTS AND LOCATIONS:
Locations (219):
- United States (43):
  - Research Site, Glendale, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Covina, California
  - Research Site, Fountain Valley, California
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, San Francisco, California
  - Research Site, Aurora, Colorado
  - Research Site, Denver, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Miami, Florida
  - Research Site, Plantation, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Murray, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Bloomfield Hills, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Omaha, Nebraska
  - Research Site, Midland Park, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Summerville, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, Galveston, Texas
  - Research Site, Mesquite, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Seattle, Washington
- Argentina (5):
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Quilmes
  - Research Site, Rosario
  - Research Site, San Miguel
- Australia (7):
  - Research Site, Clayton
  - Research Site, Kogarah
  - Research Site, Malvern
  - Research Site, Melbourne
  - Research Site, Mitcham
  - Research Site, Westmead
  - Research Site, Woolloongabba
- Austria (5):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Sankt Pölten
  - Research Site, Vienna
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Liège
- Brazil (5):
  - Research Site, Belo Horizonte
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São Paulo
- Research Site, Sofia, Bulgaria
- Canada (4):
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Toronto, Ontario
- Chile (2):
  - Research Site, Osorno
  - Research Site, Santiago
- China (20):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dongguan
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Heilongjiang
  - Research Site, Jinan
  - Research Site, Kunming
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Zhuzhou
- Colombia (3):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Chía
- Denmark (2):
  - Research Site, Aarhus
  - Research Site, Copenhagen
- France (12):
  - Research Site, Bois-Guillaume
  - Research Site, Bordeaux
  - Research Site, Chambray-lès-Tours
  - Research Site, Dijon
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Montivilliers
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Toulouse
- Germany (14):
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Dresden
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Freiburg im Breisgau
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Kiel
  - Research Site, Leipzig
  - Research Site, Mainz
  - Research Site, Marburg
  - Research Site, Regensburg
  - Research Site, Wuppertal
- Research Site, Athens, Greece
- Italy (9):
  - Research Site, Brescia
  - Research Site, Cona
  - Research Site, Florence
  - Research Site, Marche
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, Rome
- Japan (17):
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Kanazawa
  - Research Site, Kita-gun
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Okayama
  - Research Site, Omura-shi
  - Research Site, Ono
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Suita
  - Research Site, tabashi City
  - Research Site, Wakayama
  - Research Site, Yokohama
  - Research Site, Yotsukaido-shi
- Mexico (6):
  - Research Site, Cuernavaca
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, San Luis Potosí City
  - Research Site, Veracruz
  - Research Site, Zapopan
- Netherlands (4):
  - Research Site, Amsterdam
  - Research Site, Breda
  - Research Site, Nijmegen
  - Research Site, Rotterdam
- New Zealand (2):
  - Research Site, Hamilton
  - Research Site, Papatoetoe
- Philippines (3):
  - Research Site, Iloilo City
  - Research Site, Lipa
  - Research Site, Manila
- Poland (8):
  - Research Site, Gdynia
  - Research Site, Katowice
  - Research Site, Kielce
  - Research Site, Olsztyn
  - Research Site, Ossy
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Warsaw
- Portugal (4):
  - Research Site, Braga
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Porto
- Romania (4):
  - Research Site, Bucharest
  - Research Site, Craiova
  - Research Site, Iași
  - Research Site, Târgu Mureş
- Serbia (2):
  - Research Site, Belgrade
  - Research Site, Kragujevac
- Slovakia (3):
  - Research Site, Košice
  - Research Site, Piešťany
  - Research Site, Svidník
- South Africa (2):
  - Research Site, Cape Town
  - Research Site, Johannesburg
- Research Site, Seoul, South Korea
- Spain (12):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Castellon
  - Research Site, Granada
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Salamanca
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Vigo
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Khlong Luang
  - Research Site, Khon Kaen
- Turkey (Türkiye) (4):
  - Research Site, Istanbul
  - Research Site, Karşıyaka
  - Research Site, Kayseri
  - Research Site, Samsun
- United Kingdom (4):
  - Research Site, Cambridge
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/